CLINICAL TRIAL: NCT02511691
Title: PET/MRI Imaging of Glutamate Release in the Brain of Healthy Controls
Brief Title: PET/MRI Imaging of Glutamate Release in the Brain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enough data for a publication, decision of Sponsor-PI
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK ZH 2014-0441
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Healthy
MeSH Terms: interventions — PSS232

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-PSS232 (Other): Subjects receive baseline PET with 18F-PSS232 and stimulation PET with 18F-PSS232 after medical challenge with N-acetylcystein
  Interventions: Drug: 18F-PSS232

INTERVENTIONS:
Drug: 18F-PSS232 — Diagnostic PET Tracer
  Other Names: 18FABP

SUMMARY:
Based on PET (18-PSS232) and MRI, glutamate release after N-acetylcystein challenge will be monitored in human brains.

DETAILED DESCRIPTION:
Diagnostic trial with quantification of glutamate release in PET/MR.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer

Exclusion Criteria:

* smoker
* drug addiction
* significant neurological or psychiatric conditions

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03-03 (Actual); Study Completion 2016-03-03 (Actual)

PRIMARY OUTCOMES:
Difference of Binding Potentials of 18F-PSS232 in different brain regions between Baseline PET and PET after medical challenge | Baseline PET and PET after medical challenge will be scanned within 3 months
  for details, please see Innis: Journal of Cerebral Blood Flow & Metabolism (2007) 27, 1533-1539

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Buck, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- University Hopsital Zurich, Zurich, Switzerland